CLINICAL TRIAL: NCT03370523
Title: Epidemiology of Polipharmacy and Potential Drug-Drug Interactions in Elderly Cardiac Outpatients
Acronym: EPIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, EDA ÖZLEK, Faculty of Medicine, Department of Cardiology, M.D., Principal Investigator, Muğla Sıtkı Koçman University
Other Study IDs: MuglaSKUTRH
Record Dates: First submitted 2017-12-01; First posted 2017-12-12 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Polypharmacy; Drug-drug Interactions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention is planned in our study — No intervention is planned in our study

SUMMARY:
As the proportion of elderly population increasing over the last years, polypharmacy and drug-drug interactions (DDI) has been a common health care problem. This study will be performed to find out to prevalence of polypharmacy, inappropriate drug use and DDIs in in elderly patients presenting to a outpatient cardiology clinics.

DETAILED DESCRIPTION:
Objective:

As the proportion of elderly population increasing over the last years, polypharmacy and drug-drug interactions (DDI) has been a common health care problem. However, very limited epidemiologic data are available describing polypharmacy, potentially DDIs, and potentially inappropriate medications and their consequences in elderly Turkish patients. Therefore, this study will be performed to find out to prevalence of polypharmacy, inappropriate drug use and DDIs in elderly patients presenting to a outpatient cardiology clinics.

Methods:

The EPIC (Epidemiology of Polipharmacy and Potential Drug-Drug Interactions in Elderly Cardiac Outpatients) study will be the first large-scale, observational, real-world multicenter study to evaluate DDIs ve polypharmacy in elderly cardiac outpatients conducted in Turkey. We will enroll all consecutive patients (aged≥ 65 years) admitted to the outpatient cardiology clinics from January 30, 2018, through June 30, 2018, provided written informed consent. Approximately 5000 patients will be enrolled in this non-interventional study. All the data will be collected at one point in time and current clinical practice will be evaluated.

Results:

Patient demographics, disease characteristics, laboratory test results and medications used willl be collected by self reports and medical records. The severity of comorbid diseases will be recorded and scored according to Charlson comorbidity index (CCI) and patients will be divided into three groups: mild, with CCI scores of 1-2; moderate, with CCI scores of 3-4; and severe, with CCI scores ≥5. Polypharmacy will be defined as being on five or more medications at one time, DDIs will be checked with Lexicomp® and and potentially inappropriate medications will be defined with 2015 update of Beers criteria. Severe drug interactions will be defined with category D or X DIs.

Conclusion:

EPIC will be the first study evaluating polypharmacy, potentially inappropriate medications and DDIs in elderly cardiac outpatients in a real world clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients with aged ≥ 65 years

Exclusion Criteria:

* Patients under 65 years of age
* Patients who do not want to participate in our study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All consecutive patients older than 65 years who presented to cardiology outpatient clinics will be screened.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-07-30 (Actual); Primary Completion 2019-07-30 (Estimated); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of polypharmacy | 6 months
  Polypharmacy will be defined as being on five or more medications at one time.
Severity of comorbid diseases | 6 months
  The severity of comorbid diseases will be recorded and scored according to Charlson comorbidity index (CCI) and patients will be divided into three groups: mild, with CCI scores of 1-2; moderate, with CCI scores of 3-4; and severe, with CCI scores ≥5.
Drug-drug interactions | 6 months
  DDIs will be checked with Lexicomp®. Severe drug interactions will be defined with category D or X DIs.
Prevalence of inappropriate medications | 6 months
  Potentially inappropriate medications will be defined with 2015 update of Beers criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Nizip State Hospital, Gaziantep, Turkey (Türkiye)

REFERENCES:
- [Derived] Ozlek E, Cekic EG, Ozlek B, Cil C, Celik O, Dogan V, Basaran O, Tanik VO, Ozdemir HI, Celik Y, Kacmaz C, Simsek Z, Gunes HM, Safak O, Ozkan B, Tasar O, Onal C, Bekar L, Biteker M. Rationale, design, and methodology of the EPIC (Epidemiology of Polypharmacy and Potential Drug-Drug Interactions in Elderly Cardiac Outpatients) study. Turk Kardiyol Dern Ars. 2019 Jul;47(5):391-398. doi: 10.5543/tkda.2019.27724. PMID 31311898